CLINICAL TRIAL: NCT04164862
Title: Effectiveness of AccuVein AV400 Device Versus Ultrasound-guided Cannulation of the Great Saphenous Vein at the Ankle in Infants: A Randomized Controlled Trial
Brief Title: AccuVein AV400 Device Versus Ultrasound-guided Cannulation of the Great Saphenous Vein at the Ankle in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assistant Professor of Aneasthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00012098; 00018699 (Other: Ethics committee Alexandria University)
Record Dates: First submitted 2019-11-05; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Intravenous Cannulation
Keywords: AccuVein AV400 device; ultrasound-guided cannulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- use ACCUVEIN AV400 (Active Comparator): Device to facilitate cannulation of the great saphenous vein at the ankle in infants
  Interventions: Device: AccuVein AV400 Device Versus Ultrasound-guided Cannulation
- ULTRASOUND GUIDED CANNULATION (Active Comparator): Ultrasound cannulation of the great saphenous vein in infants
  Interventions: Device: AccuVein AV400 Device Versus Ultrasound-guided Cannulation

INTERVENTIONS:
Device: AccuVein AV400 Device Versus Ultrasound-guided Cannulation — Accuvein AV400 device versus Ultrasound guided cannulation

SUMMARY:
Establishment of venousaccess in the age group ≤12 months can be difficult and associated with repetitive punctures . Numerous techniques to facilitate peripheral venous puncture have been described such as local warming, epidermal nitrogycerine, translumination, and venous cutdown . Ultrasound guidance is reported to facilitate peripheral venous catheterisation in children and to have advantages over blind techniques, especially for challenging veins . Also The AccuVein AV400 device which detects the haemoglobin in the vessels by red and infrared light reflection and shows a vasculature map. AccuVein AV400 device (AV400) improves the success rate of intravenous cannulation in pediatric patients .

Most peripheral veins in infants are too superficial and too small for direct visualization. A promising alternative approach could be the great saphenous vein (GSV) at the level of the medial malleolus due to the adequate diameter and the relatively deep position relative to the skin.

DETAILED DESCRIPTION:
The present study is designed to investigate the practicability of ultrasound-guided vascular access versus the AccuVein AV 400 for cannulation of the great saphenous vein at the level of the medial malleoli in infants ≤12 months. The primary outcome will be the time to successful placement of catheters. Secondary outcomes included the number of attempts, the rate of failure, technique-related pain, occurrence of movements, and occurrence of complications like haematoma or local infection.

Patient and method:

A prospective, randomized study will be conducted from May 2019 till November 2019; at least 50 patients will be allocated in each group; at the Alexandria Main University Hospital after approval of the Medical Ethics Committee. Informed written consent will be obtained from the patient's parents. Infants' ≤12 months with ASA physical status I and II, undergoing elective surgery with no visible veins at the dorsum of the hands or feet will be enrolled in the study. Infants will be randomly assigned, by using a block of four randomization provided by www.randomization.com, into two groups; an AV400 group (using the AccuVein AV400 for peripheral venous insertion) and a ultrasound guided group (using the ultrasound for peripheral venous insertion). The performers of cannulation will be done by expert anesthetists, having a minimum of 5 times experience in ultra sound guided IV cannula insertion and with the AccuVein AV400 device.

Preoperatively in all infants, both medial malleolar areas will be prepared with EMLA cream , premedication with 1 mg/ kg rectal midazolam (maximum dose 15 mg) will be done at 30 minutes preoperative. Establishment of standard monitoring (SpO2, ECG, non-invasive arterial pressure) and then induction of general anaesthesia will be done via a face mask with sevoflurane FIO2 40% - O2/air and after successful induction of general anaesthesia, the EMLA tapes will be removed .Assisted ventilation via the face mask will be done until establishment of venous access either through using Acc Vein AV400 or through ultrasound guided for the great saphenous vein. On each occasion, the observer will record the time of tourniquet application, the time of successful cannulation or four skin punctures, and the number of cannulation attempts. A cannulation attempt will be defined as any backward and forward movements of the needle, regardless of whether the needle was out of the skin. Successful cannulation will be defined by the absence of tissue swelling around the puncture point after injection of 5 ml of crystalloid solution. In both groups, a maximal number of three attempts for establishment of venous access in one GSV will be performed. If the third attempt failed, the contralateral GSV will be punctured. If successful establishment of venous access in the contralateral GSV failed, the case will be counted as failure. In these cases, the external jugular vein will be used as an alternative approach for venous access. After successful establishment of venous access, the anaesthetic procedure will be continued depending on surgical requirements. Twenty-four hours after establishment of the venous access, the puncture site will be evaluated to detect possible haematoma or local infection.

ELIGIBILITY:
Inclusion Criteria:

* Infants' ≤12 months
* ASA physical status I and II
* undergoing elective surgery
* with no visible veins at the dorsum of the hands or feet

Exclusion Criteria:

• REFUSAL

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
the time to successful placement of catheters | "Through operation completion, average of 2 hours"
  the time to successful placement of catheters

SECONDARY OUTCOMES:
the number of attempts | "Through operation completion, average of 2 hours"
  attempts for successful cannulation
, technique-related pain, occurrence of movements, and occurrence of complications . | "Through operation completion, average of 2 hours"
  complications like haematoma or local infection.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Zayed, Ass.Prof., Principal Investigator — Alexandria University; yasser Osman, Ass. Prof., Principal Investigator — Alexandria University
Locations (1):
- Rehab A.Zayed, Alexandria, Egypt